CLINICAL TRIAL: NCT07050420
Title: The Effectiveness of Child Abuse and Neglect Education Given to Nurses Working in Pediatric Clinics on Their Awareness Levels: A Randomized Controlled Study
Brief Title: Child Abuse Training Impact on Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, SEDA TEK SEVİNDİK, PhD, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IstanbulMedeniyetU
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Child Abuse
Keywords: Pediatric clinics; nursing; child abuse; child neglect; awareness

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Clinic Nurses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group Nurses (Active Comparator): Nurses who will receive training on child abuse and neglect
  Interventions: Other: Training
- Comparison Group Nurses (No Intervention): Nurses who will not receive training in child abuse and neglect

INTERVENTIONS:
Other: Training — Education on Child Abuse and Neglect
  Arms: Training Group Nurses

SUMMARY:
This study aims to determine the effect of the training given to nurses working in pediatric clinics on child abuse and neglect on the awareness levels of nurses regarding child abuse and neglect.

DETAILED DESCRIPTION:
* H0: Education given to nurses working in pediatric clinics about child abuse and neglect has no effect on nurses' awareness of child abuse and neglect.
* H1: Education given to nurses working in pediatric clinics about child abuse and neglect has an effect on nurses' awareness of child abuse and neglect.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate voluntarily in the study and signing the informed consent form.
* Being a nurse working in the pediatric clinics and pediatric emergency department at Cukurova University Balcali Hospital Health Application and Research Center during the data collection dates of the study.

Exclusion Criteria:

* Nurses who do not want to participate in the study or leave the process will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-17 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Scale Form for Diagnosing Signs and Risks of Child Abuse and Neglect | 3 times; a week before training, a week after training, 1 month after training
  There are 6 subscales in the scale form for diagnosing the symptoms and risks of child abuse and neglect. These are; Physical symptoms of abuse on children (19 items), Behavioral symptoms of child abuse (15 items), Symptoms of neglect on children (7 items), Characteristics of parents prone to abuse and neglect (13 items), Characteristics of children prone to abuse and neglect (5 items), Familial characteristics in child abuse and neglect (8 items). Likert-type scale for determining the knowledge levels of nurses and midwives in diagnosing the symptoms and risks of child abuse and neglect. A score average approaching 5 indicates that they are knowledgeable about the signs and risks of child abuse and neglect, and a score away from 3 indicates that they are not knowledgeable about the signs and risks of child abuse and neglect. A subject who answers all items of the scale form correctly is expected to receive a full score of 335.

IPD SHARING:
Plan to Share IPD: No